CLINICAL TRIAL: NCT02432573
Title: Timing of Morning Rounds for Postpartum Hospitalized Women: A Randomized Controlled Quality Improvement Trial
Brief Title: Timing of Morning Rounds for Postpartum Hospitalized Women
Acronym: PP rounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robyn Roberts, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSC-MS-15-0245
Record Dates: First submitted 2015-04-09; First posted 2015-05-04 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Physician Rounds; Postpartum
Keywords: timing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Postpartum patients that receive physician rounding at current time
- Delayed rounding (Experimental): Postpartum patients that receive physician rounding at a delayed time
  Interventions: Behavioral: Delayed rounds

INTERVENTIONS:
Behavioral: Delayed rounds
  Arms: Delayed rounding

SUMMARY:
In postpartum hospitalized women, does delayed morning rounding improve patient satisfaction?

DETAILED DESCRIPTION:
OBJECTIVE To investigate the timing of physician rounds on patient satisfaction

STUDY DESIGN Randomized, controlled, quality improvement trial

OUTCOMES Primary: score on Hospital Consumer Assessment of Healthcare Provers and Systems (HCAPS) survey

Secondary: score on Edinburgh Postnatal Depression Scale

ELIGIBILITY:
Inclusion Criteria:

* Delivered between 0600 and 0000
* Admitted to Memorial Hermann postpartum unit
* Patient managed by the University of Texas Physicians Group and/or obstetrics-gynecology residents

Exclusion Criteria:

- None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
score on Hospital Consumer Assessment of Healthcare Provers and Systems (HCAPS) survey | 2 months
  Patient will be give a modified version of the validated HCAPS survey at discharge from the hospital to assess patient satisfaction and the scores will be compared between the 2 groups.

SECONDARY OUTCOMES:
score on Edinburgh Postnatal Depression Scale | 2 months
  Patient will be given this questionnaire at discharge from the hospital to assess risk for postpartum depression and the scores will be compared between the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn P Roberts, MD, Principal Investigator — University of Texas
Locations (1):
- Texas Medical Center, Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Roberts RP, Blackwell SC, Brown KM, Pedroza C, Sibai BM, Tyson JE. Early Compared With Delayed Physician Rounds on Patient Satisfaction of Postpartum Women: A Randomized Controlled Trial. Obstet Gynecol. 2016 Aug;128(2):381-386. doi: 10.1097/AOG.0000000000001528. PMID 27400002